CLINICAL TRIAL: NCT07102173
Title: Management Protocol for Comparison of Loco-regional Analgesic Techniques in Patients Undergoing Video Assisted Thoracoscopic Surgery (VATS)
Brief Title: Comparison of Loco-regional Analgesic Techniques in Patients Undergoing Video Assisted Thoracoscopic Surgery (VATS)
Acronym: PRoGEVATS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ASST Sette Laghi (Other)
Responsible Party: Principal Investigator, Luca Guzzetti, MD, Ospedale di Circolo - Fondazione Macchi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 209/2024
Record Dates: First submitted 2025-07-14; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Loco-regional Anesthesia
Keywords: VATS; post-operative analgesia; loco-regional anesthesia; ESPB; Intercostal nerve block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intercostal nerve block (Active Comparator): Performed by the surgeon intraoperatively before final lung re-expansion, involving the administration of 20 mL of 0.5% levobupivacaine using a 27G needle into the subpleural space of the thoracotomy access site and adjacent intercostal spaces.
  Interventions: Procedure: Intercostal nerve block
- Ultrasound-guided ESPB (Active Comparator): Performed by an anesthesiologist under surgical asepsis with the patient in a seated position. After identifying the target transverse process, a linear ultrasound probe is placed sagittally approximately 2 cm from the midline. The needle (22G, 50 mm) is inserted in-plane in a cranio-caudal direction until contacting the transverse process. After confirming proper injection by observing anesthetic spread between the erector spinae muscle and transverse process, a total of 30 mL of 0.375% ropivacaine is administered.
  Interventions: Procedure: Ultrasound-guided ESPB

INTERVENTIONS:
Procedure: Intercostal nerve block — Before final lung re-expansion, involving the administration of 20 mL of 0.5% levobupivacaine using a 27G needle into the subpleural space of the thoracotomy access site and adjacent intercostal spaces.
  Arms: Intercostal nerve block
Procedure: Ultrasound-guided ESPB — After identifying the target transverse process, a linear ultrasound probe is placed sagittally approximately 2 cm from the midline. The needle (22G, 50 mm) is inserted in-plane in a cranio-caudal direction until contacting the transverse process. After confirming proper injection by observing anesthetic spread between the erector spinae muscle and transverse process, a total of 30 mL of 0.375% ropivacaine is administered.
  Arms: Ultrasound-guided ESPB

SUMMARY:
This study aims to compare two loco-regional analgesic techniques:

1. Intercostal nerve block: Performed by the surgeon intraoperatively before final lung re-expansion, involving the administration of 20 mL of 0.5% levobupivacaine using a 27G needle into the subpleural space of the thoracotomy access site and adjacent intercostal spaces.
2. Ultrasound-guided ESPB: Performed by an anesthesiologist under surgical asepsis with the patient in a seated position. After identifying the target transverse process, a linear ultrasound probe is placed sagittally approximately 2 cm from the midline. The needle (22G, 50 mm) is inserted in-plane in a cranio-caudal direction until contacting the transverse process. After confirming proper injection by observing anesthetic spread between the erector spinae muscle and transverse process, a total of 30 mL of 0.375% ropivacaine is administered.

This protocol is intended for patients undergoing video-assisted thoracoscopic surgery (VATS) for pneumonectomies, lobectomies, wedge resections, and bullectomies.

Primary Endpoint:QoR Score at 24 hours (validated questionnaires. Secondary Endpoints: Intraoperative NOL, QoR at 48-72 hours, opioid consumption at 12-24-48 hours, NLR at 24 hours, CPSP incidence at 3 months.

DETAILED DESCRIPTION:
Video-assisted thoracoscopic surgery (VATS) is a minimally invasive procedure that offers numerous advantages over traditional thoracotomy, including reduced surgical stress, lower postoperative pain, improved postoperative pulmonary function, reduced mortality, and shorter hospital stays.

Although VATS is less painful than open surgery, patients may still experience significant postoperative pain. Therefore, effective pain management is crucial to reducing postoperative complications and preventing acute postoperative pain from progressing to chronic pain.

Thoracic epidural analgesia and thoracic paravertebral blocks provide adequate pain control for thoracic surgery but may be associated with complications that can prolong hospital stays and increase morbidity.

Thus, recent trends favor less invasive regional analgesic techniques combined with systemic analgesia. Systemic analgesia follows a multimodal approach, incorporating intravenous medications such as acetaminophen, NSAIDs, lidocaine, and α2-adrenergic agonists.

Recent PROSPECT (PROcedure SPECific Postoperative Pain ManagemenT) guidelines recommend the erector spinae plane block (ESP) or paravertebral block (PVB) for postoperative analgesia following VATS.

Given the variety of available techniques, it is essential to determine the most effective analgesic strategy for postoperative pain management in VATS. Additionally, a standardized method for assessing both acute and chronic postoperative pain is necessary.

Furthermore, adopting an Enhanced Recovery After Surgery (ERAS) approach in thoracic surgery may be beneficial. ERAS is a perioperative care program involving multiple evidence-based interventions aimed at reducing surgical stress and accelerating patient recovery. Postoperative recovery is influenced by several factors, including the patient's general health status, anesthesia, and surgical techniques. One critical aspect of postoperative recovery assessment is the patient;s perception of their recovery quality, encompassing well-being, overall quality of life, and recovery from anesthesia. One of the most widely used tools for assessing perceived recovery quality is the Quality of Recovery-40 (QoR-40) questionnaire, developed by Myles in 2020. It evaluates five dimensions: pain, physical comfort, physical independence, emotional state, and psychological support. A shorter 15-item version (QoR-15) was later developed, which maintains good validity, reliability, and feasibility, as most patients can complete it in under three minutes.

Intraoperatively, technological advancements have led to the development of highly sophisticated analgesic monitoring tools. The Nociception Level Index (NOL®) is an innovative technology developed by Medasense Biometrics Ltd. that objectively measures nociception by analyzing multiple physiological parameters through artificial intelligence algorithms. A non-invasive fingertip probe with four sensors (photoplethysmography, galvanic skin response, peripheral temperature, and accelerometry) extracts multiple pain- related physiological signals. The algorithms analyze the data in real-time to identify the patient's pain patterns, translating them into a numerical scale. This device enables precise nociception monitoring in anesthetized patients, allowing for personalized analgesic treatment.

Postoperative pain remains a challenge in patients undergoing VATS, as inadequate acute pain control increases the risk of immediate complications and contributes to the development of chronic pain, leading to prolonged postoperative opioid use.

Balancing the efficacy of loco-regional analgesic techniques with their invasiveness and risk of procedural complications is essential. Recent literature suggests that both intraoperative intercostal nerve blocks and ultrasound-guided erector spinae plane blocks (ESPB) provide effective analgesia while being clinically safe and technically simple.

ESPB, in particular, allows anesthetic spread to both dorsal and ventral spinal nerve branches, covering approximately four dermatomes above and below the injection site.

Few comparative studies exist between these two techniques, indicating non-inferiority in terms of postoperative pain scores (NRS) and opioid consumption at 48 hours. However, further research is needed to assess intraoperative efficacy, postoperative complications, quality of recovery, and chronic pain development in patients receiving these techniques.

Chronic post-surgical pain (CPSP) is defined by the International Classification of Diseases (ICD-11) as "pain that develops or increases in intensity following a surgical procedure and persists beyond the healing process for at least three months postoperatively; it is localized to the surgical area or the nerve distribution area in that region; other identifiable causes of pain must be excluded, and it may present with neuropathic characteristics." Given that CPSP affects 10%-50% of surgical patients, even a modest reduction in its prevalence could significantly improve many patients; quality of life. Inflammation plays a key role in acute pain generation and in mediating the transition from acute to chronic postoperative pain. The postoperative release of pro-inflammatory cytokines and chemokines contributes to peripheral and central sensitization, which are critical mechanisms underlying CPSP. Elevated absolute neutrophil counts, high neutrophil-to-lymphocyte ratio (NLR), or low absolute lymphocyte counts postoperatively have been associated with an increased risk of CPSP. A modified NLR ratio (postoperative/preoperative) ≥ 5 has been significantly correlated with CPSP in orthopedic procedures, shoulder arthroscopy, dental surgery, and laparoscopic cholecystectomy.

However, its correlation with CPSP in thoracic surgery remains unclear.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Signed informed consent
* Elective unilateral surgery

Exclusion Criteria:

* Minor patients
* BMI > 40
* Unstable neurological disorders
* Known allergy to acetaminophen and NSAIDs
* Chronic renal failure (stage > 4, whith GFR between 29 and 15 mL/min)
* Patient refusal
* Chronic use of NSAIDs and opioids in the 3 months prior to surgery
* Contraindications to peripheral block (infection al the insertion site, allergy to local anesthetics, severe coagulation disorders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
QoR Score at Day 1 | From end surgery to Day 1 after surgery

SECONDARY OUTCOMES:
Intraoperative NOL (Nociception Level Index®) | From start to end surgery
  NOL (Nociception Level) is the technology and index to objectively quantify a patient's physiological pain response (nociception). The Nociception Level index (NOL™) is a multiparameter index, based on artificial intelligence for the monitoring of nociception during anesthesia. We record the NOL number to assess nociceptive stimulation during surgery.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code